CLINICAL TRIAL: NCT03707418
Title: A Randomized Study Comparing Bivalirudin vs Heparin in Patients With Extracorporeal Membrane Oxygenator (ECMO) Support
Brief Title: Bivalirudin vs Heparin in ECMO Patients
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: unable to secure funding
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00176475
Record Dates: First submitted 2018-10-11; First posted 2018-10-16 (Actual); Last update posted 2021-01-19 (Actual); Status verified 2020-04

CONDITIONS: Extracorporeal Membrane Oxygenation Complication
MeSH Terms: interventions — Heparin; bivalirudin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Bivalirudin Injection (Angiomax) (Active Comparator): This arm will receive intravenous Bivalirudin for ECMO anticoagulation for the extent of ECMO support or 7 days whichever comes first
  Interventions: Drug: Bivalirudin Injection [Angiomax]
- Heparin Sodium (Active Comparator): This arm will receive intravenous Heparin Sodium for ECMO anticoagulation for the extent of ECMO support or 7 days whichever comes first
  Interventions: Drug: Heparin Sodium

INTERVENTIONS:
Drug: Heparin Sodium — Intravenous Heparin titrated to Partial ThromboplastinTime (PTT) levels
  Arms: Heparin Sodium
Drug: Bivalirudin Injection [Angiomax] — Intravenous Bivalirudin titrated to Activated Clotting Time (ACT) levels
  Arms: Bivalirudin Injection (Angiomax)

SUMMARY:
This is an open label, randomized study comparing the clinical outcomes of unfractionated Heparin and Bivalirudin for anticoagulation in adult subjects requiring ECMO support.

DETAILED DESCRIPTION:
This open label randomized study will compare the clinical outcomes of patients on ECMO who are anticoagulated with Heparin and Bivalirudin. Patients will be anticoagulated with a heparin bolus at the commencement of ECMO per standard of care, as there will be insufficient time to randomize these frequently emergent patients. Consent for the study will be obtained from a legally authorized representative Prior to starting a continuous infusion of maintenance anticoagulation, patients will be randomized to bivalirudin or heparin. Outcome measures are bleeding, thrombosis, development of Heparin Induced thrombocytopenia, number of cross-overs between the two research arms, circuit failures, decannulation, deaths and discharges from hospital.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients on veno-arterial (VA) or veno-venous (VV)ECMO

Exclusion Criteria:

* Patient or surrogate decision makers cannot provide informed consent.
* Patients who have intolerance to either heparin or bivalirudin
* Patients who received any form of thrombolytic therapy within the past 30 days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-04 (Estimated); Primary Completion 2021-06 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
Number of heparin-induced thrombocytopenia (HIT) events | 30 days
  This will be assessed by serum platelet factor 4 antibody level
Number of Cross-overs between arms | 30 days
  This will be assessed by number of cross over of patients from one arm to the other anti-coagulation arm for any particular clinical reason.
  Crossover patients will remain in the study and we will continue to collect protocol driven data. These patients will be analyzed separately from those with no cross-over.
Number of circuit failures requiring a circuit exchange | 30 days
  Will be determined by total number of circuit exchanges needed in ECMO circuit due to thrombosis. Circuit exchanges may be done due to lack of adequate gas exchange or increased resistance pre and post oxygenator >50mmHg, circuit thrombosis or failure requiring emergent decannulation
Thrombotic events | 30 days
  Collect number of thrombotic events, defined as any of the following events; embolic strokes, embolic end-organ ischemia, embolic ischemia to limbs, deep vein thrombosis or venous thromboembolism, Oxygenator effectiveness measured by resistance, Alveolar-arterial oxygen gradient and carbon dioxide elimination
Bleeding events | 30 days
  Will be assessed by the total number of one or more of the following: Chest tube output of blood, number of take-backs to operating room for bleeding, number of Hemorrhagic strokes, Gastrointestinal bleeding, Retroperitoneal hemorrhage, number of cessations of anticoagulation for refractory bleeding and any use of antifibrinolytics or factor VII
Renal failure | 30 days
  Defined as initiation of renal replacement therapy for kidney injury that develops on ECMO or increase in serum creatinine by more than 2 times its baseline or decrease in Glomerular Filtration Rate by more than 50% or urine output less than 0.3 mL/kg/hr. We will determine the number of patients with renal failure
Number of Transfusions | 30 days
  This will be assessed by any of the following: number of utilizations of packed red blood cells and utilization of fresh frozen plasma, utilization of platelets, utilization of cryoprecipitate, utilization of anti-thrombin III, utilization of factor VII, utilization of prothrombin complex concentrate
Number of emergent decannulations | 30 days
  This will be assessed by the number of times patient is separated from ECMO
Number of patients surviving to discharge | 30 days
  This will be assessed by the number of patients in each arm who survive to discharge

CONTACTS AND LOCATIONS:
Overall Officials: Glenn Whitman, M.D., Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Hasegawa D, Sato R, Prasitlumkum N, Nishida K, Keaton B, Acquah SO, Im Lee Y. Comparison of Bivalirudin Versus Heparin for Anticoagulation During Extracorporeal Membrane Oxygenation. ASAIO J. 2023 Apr 1;69(4):396-401. doi: 10.1097/MAT.0000000000001814. Epub 2022 Apr 10. PMID 36194483